CLINICAL TRIAL: NCT01629043
Title: Parkinson's Foundation Quality Improvement Initiative
Acronym: PF-QII
Status: Completed | Type: Observational
Sponsor: National Parkinson Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Parkinson's Foundation-QII
Record Dates: First submitted 2012-06-25; First posted 2012-06-27 (Estimated); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's; Quality of Care; Improvement; Mobility; Cognition; Caregiver burden; Center difference
MeSH Terms: conditions — Parkinson Disease; Caregiver Burden

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In a recent study it was found that neurologist care for Parkinson's provides a 20% reduction in nursing home placement, hip fracture, and death (Willis 2011). However, as the authors recognized, the investigators don't know what it is about expert care that delivers this benefit. The Parkinson's Foundation's Quality Improvement Initiative was designed to identify the components of great care that yield great outcomes. By capturing demographics, clinical interventions and outcomes over time from multiple centers across the U.S, Canada and internationally, the best care practices from different clinics and different healthcare systems will be analyzed.

DETAILED DESCRIPTION:
In a recent study it was found that neurologist care for Parkinson's provides a 20% reduction in nursing home placement, hip fracture, and death (Willis 2011). However, as the authors recognized, we don't know what it is about expert care that delivers this benefit. The Parkinson's Foundation's Quality Improvement Initiative was designed to identify the components of great care that yield great outcomes. By capturing demographics, clinical interventions and outcomes over time from multiple centers across the U.S, Canada and internationally, the best care practices for improving care, survival, and quality of life from different clinics and different healthcare systems will be analyzed.

The Parkinson's Foundation's QII contains demographic data, information about the patient's Parkinson's disease and other comorbid illness, patient assessments of Parkinson's related physical, emotional and cognitive disability and clinician tests of mobility, memory and cognition. It also includes data on the burden of the disease on caregivers. The tests and questionnaire instruments are currently in regular use in clinical practice. The intent of the registry is not to evaluate the instruments themselves but to collect essential data from previously validated tools.

Registry data will be used to study the relationship between treatment and clinical symptoms of patients with Parkinson's. It will also be used to evaluate and improve care of patients at participating Centers. Through presentation and publication of results, it is hoped that improvement will become more widespread. Important benefits provided by such a Registry may ultimately be to:

* Determine the long term effects of Parkinson's disease and related conditions on quality of life;
* Generate regular reports for Centers including descriptions of their Parkinson's patient populations, treatments utilized at the Center and trends in their patients' outcomes over time;
* Describe differences in current practice across Centers in the care of Parkinson's patients;
* Identify patients who may be candidates for participation in trials of new medications;
* Facilitate or initiate quality improvement efforts intended to enhance survival and/or improve quality of life for Parkinson's disease patients; and
* Publish and otherwise disseminate findings related to most effective treatments to encourage rapid adoption of "best practices."

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic Parkinson's disease receiving medical care for the diagnosis of idiopathic Parkinson's disease at any of the participating Centers.

Exclusion Criteria:

Patients who are not willing or won't be able to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any person who receives medical care for the diagnosis of idiopathic Parkinson's disease at any of the participating Centers is eligible to participate in the Registry. There are no limitations for participation based on age, disease severity or presence of cognitive impairments.
Sampling Method: Probability Sample
Enrollment: 13000 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2023-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Davis, MD, Study Chair — Vanderbilt University Medical Center; Adolfo Ramirez-Zamora, MD, Study Chair — University of Florida; Kelly Lyons, PhD, Study Chair — University of Kansas Medical Center
Locations (24):
- United States (18):
  - Barrow Neurological Institute - Muhammad Ali Parkinson Center, Phoenix, Arizona
  - Parkinson's Institute and Clinical Center, Sunnyvale, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida Parkinson's Disease and Movement Disorders Center, Gainesville, Florida
  - University of Miami Parkinson's Disease and Movement Disorders Center, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Northwestern University Parkinson's Disease and Movement Disorders Center, Chicago, Illinois
  - University of Kansas Medical Center Parkinson's Disease and Movement Disorder Center, Kansas City, Kansas
  - Johns Hopkins Parkinson's Disease and Movement Disorder Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center Parkinson's Disease Movement Disorder Center, Boston, Massachusetts
  - Struthers Parkinson Center, Golden Valley, Minnesota
  - NYU Langone Medical Center, New York, New York
  - Mount Sinai School of Medicine Parkinson and movement Disorders Center, New York, New York
  - Oregon Health and Science University Parkinson Center, Portland, Oregon
  - University of Pennsylvania Parkinson's Disease and Movement Disorder Center, Philadelphia, Pennsylvania
  - The Vanderbilt Parkinson Disease Center, Nashville, Tennessee
  - Baylor College of Medicine Parkinson Disease Center and Movement Disorders Clinic, Houston, Texas
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - Centre for Movement Disorders, Markham, Ontario
  - Toronto Western Hospital Movement Disorders Center, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Parkinson Center Nijmegen at Radboud University Nijmegen Medical Center, Nijmegen, Netherlands

REFERENCES:
- [Background] Okun MS, Siderowf A, Nutt JG, O'Conner GT, Bloem BR, Olmstead EM, Guttman M, Simuni T, Cheng E, Cohen EV, Parashos S, Marsh L, Malaty IA, Giladi N, Schmidt P, Oberdorf J. Piloting the NPF data-driven quality improvement initiative. Parkinsonism Relat Disord. 2010 Sep;16(8):517-21. doi: 10.1016/j.parkreldis.2010.06.005. Epub 2010 Jul 6. PMID 20609611